CLINICAL TRIAL: NCT05270551
Title: The Effect of Accelerated Rehabilitation After Anterior Cruciate Ligament Reconstruction With and Without Suture Tape Reinforcement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACL Recon. rehabilitation
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: ACL Injury
Keywords: Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Without augmentation
  Interventions: Procedure: ACL Reconstruction
- Group 2 (Active Comparator): With augmentation
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: ACL Reconstruction — All participants will do ACL reconstruction with and without Augmentation and will receive Accelerated rehabilitation program

SUMMARY:
The aim of our study is to evaluate the effect of accelerated rehabilitation post ACL reconstruction with and without augmentation on graft healing and return to normal activity clinically by scoring system and radiologically.

DETAILED DESCRIPTION:
ACL reconstruction is the most commonly performed knee ligament reconstruction and employs a variety of surgical techniques. However, despite high success rates, it is still challenged by residual laxity and graft rupture.

While the majority of patients who undergo ACLR will have good to excellent results, a subset of patients is at a higher risk for graft failure. For those that require revision surgery, the second operation often fails. Anterior cruciate ligament injuries account for 50% of knee ligament injuries for high school-aged adults.

The most commonly used autografts for ACLR are the hamstring tendons (HT) and the bone-patellar tendon-bone (BPTB). However, questions remain about how patients with either an HT or a BPTB autograft recover knee muscle strength postoperatively.

To help address and prevent future ACL failures, new repair and reconstruction techniques have been employed that incorporate suture augmentation. The goal of augmentation is to protect the newly repaired or reconstructed ligament during rehabilitation.

Despite advances in anterior cruciate ligament (ACL) reconstruction surgical techniques and rehabilitation, recent studies report that between 20% to 50% of those with ACL reconstruction do not return to the same sports after surgery and 10% to 70% of those who resume preinjury sports participate at a reduced level or with significant functional impairments.

Anecdotal evidence from patient report and clinical observation suggests that an inability to return to sports after ACL reconstruction can be partially attributed to a fear of reinjuring the knee.

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 50 years old.
* With or without meniscal injury.
* Isolated ACL injury without any other ligament injury.
* Recent and chronic injury.

Exclusion Criteria:

* Multiligament injury.
* Deformed knee (Genu varus or valgus).
* Previous ACL reconstruction or repair.
* Older than 50 years old and younger than 15 years old.
* Failed ACL reconstruction or repair -

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 1 year follow up
  Tegner Lysholm scores, which assesses activity levels
Clinical outcome | 1 year follow up
  International Knee Documentation Committee (IKDC) scores which assesses symptoms and function in daily living activities

SECONDARY OUTCOMES:
Radiological outcome | 6 months follow up
  Magnetic resonance imaging (MRI) to assess graft healing, ACL tear and graft loosening

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel Hamid, Professor, Study Chair — Mohamad Mohamed Abdel-Hamid Morsy; Hatem Galal El-Din Zaki, Professor, Principal Investigator — Hatem Galal El-Din Zaki; Mohamed Abd El-Radi, Lecturer, Study Director — Mohamed Abd El-Radi Abd El-Salam

REFERENCES:
- [Background] Schlumberger M, Schuster P, Schulz M, Immendorfer M, Mayer P, Bartholoma J, Richter J. Traumatic graft rupture after primary and revision anterior cruciate ligament reconstruction: retrospective analysis of incidence and risk factors in 2915 cases. Knee Surg Sports Traumatol Arthrosc. 2017 May;25(5):1535-1541. doi: 10.1007/s00167-015-3699-0. Epub 2015 Sep 26. PMID 26410092
- [Background] Riediger MD, Stride D, Coke SE, Kurz AZ, Duong A, Ayeni OR. ACL Reconstruction with Augmentation: a Scoping Review. Curr Rev Musculoskelet Med. 2019 Jun;12(2):166-172. doi: 10.1007/s12178-019-09548-4. PMID 30945237
- [Background] Cristiani R, Mikkelsen C, Wange P, Olsson D, Stalman A, Engstrom B. Autograft type affects muscle strength and hop performance after ACL reconstruction. A randomised controlled trial comparing patellar tendon and hamstring tendon autografts with standard or accelerated rehabilitation. Knee Surg Sports Traumatol Arthrosc. 2021 Sep;29(9):3025-3036. doi: 10.1007/s00167-020-06334-5. Epub 2020 Oct 31. PMID 33128587
- [Background] Smith PA, Bley JA. Allograft Anterior Cruciate Ligament Reconstruction Utilizing Internal Brace Augmentation. Arthrosc Tech. 2016 Oct 10;5(5):e1143-e1147. doi: 10.1016/j.eats.2016.06.007. eCollection 2016 Oct. PMID 28224069
- [Background] Chmielewski TL, Jones D, Day T, Tillman SM, Lentz TA, George SZ. The association of pain and fear of movement/reinjury with function during anterior cruciate ligament reconstruction rehabilitation. J Orthop Sports Phys Ther. 2008 Dec;38(12):746-53. doi: 10.2519/jospt.2008.2887. PMID 19047767
- [Background] Beynnon BD, Johnson RJ, Abate JA, Fleming BC, Nichols CE. Treatment of anterior cruciate ligament injuries, part 2. Am J Sports Med. 2005 Nov;33(11):1751-67. doi: 10.1177/0363546505279922. PMID 16230470
- [Background] Dean AG. OpenEpi: open source epidemiologic statistics for public health, version 2.3. 1. http://www. openepi. com. 2010.